CLINICAL TRIAL: NCT07085741
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (MAGNET System, DI Biofragmentable) to Achieve Duodeno-Ileostomy Diversion in Adults With Obesity and Type 2 Diabetes Mellitus: MAGNET 2 Study
Brief Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System in Mexico
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-002
Record Dates: First submitted 2025-04-08; First posted 2025-07-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter study enrolling up to 25 subjects at up to 3 study centers in Mexico
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAGNET System, DI Biofragmentable (Experimental): GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (MAGNET System, DI Biofragmentable)
  Interventions: Device: MAGNET System, DI Biofragmentable

INTERVENTIONS:
Device: MAGNET System, DI Biofragmentable — Anastomoses achieved by magnetic compression.

SUMMARY:
The purpose of this clinical research study is to evaluate the feasibility / performance, safety and initial efficacy of the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (MAGNET System, DI Biofragmentable) for creation of a side-to-side anastomosis duodeno-ileostomy in obese adults.

DETAILED DESCRIPTION:
The purpose of this clinical research study is to evaluate the feasibility/performance, safety and initial efficacy of the GT Metabolic Solutions DI Biofragmentable Magnetic Anastomosis System (MAGNET System, DI Biofragmentable) for creation of a side-to-side anastomosis duodeno-ileostomy in obese adults. This partial diversion of intestinal contents from duodenum to the ileum is intended to facilitate weight management/loss in obese adults with type 2 diabetes mellitus (T2DM) and improve metabolic outcomes in obese adults with type 2 diabetes mellitus (T2DM). Side-by side- anastomoses are currently created by sutures, staples, and anastomotic compression devices. A predicate procedure is the single-anastomosis duodeno- ileostomy (SADI) procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age, inclusive, at the time of informed consent
2. BMI 30-34.9 kg/m2
3. Type 2 Diabetes Mellitus (T2DM; defined as HbA1c 6.5%), without previous sleeve gastrectomy, and without plan to perform a concurrent sleeve gastrectomy.
4. Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for the duration of the study
5. If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for the duration of the study
6. Willing and able to comply with protocol requirements

Exclusion Criteria:

1. Type 1 diabetes
2. Use of injectable insulin
3. Uncontrolled T2DM
4. Previous sleeve gastrectomy procedure or plan to perform a sleeve gastrectomy with the duodeno-ileal anastomosis procedure
5. Uncontrolled hypertension, dyslipidemia or sleep apnea
6. Prior intestinal, colonic or duodenal surgery, other than bariatric
7. Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contra-indicate the procedure, including scarring and abnormal anatomy.
8. Refractory gastro-esophageal reflux disease (GERD)
9. Barrett's disease
10. Helicobacter pylori positive and/or active ulcer disease
11. Large hiatal hernia
12. Inflammatory bowel or colonic diverticulitis disease
13. Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques.
14. Implantable pacemaker or defibrillator
15. Psychiatric disorder, except well-controlled depression with medication for >6 months
16. History of substance abuse
17. Woman who is either pregnant or breast feeding
18. Woman of childbearing potential who does not agree to use an effective method of contraception.
19. Any comorbidity or current status of subject's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the subject medically unfit for the procedure, including any significant congenital or acquired anomalies of the GI tract at or distal to the placement of the magnets.
20. Unhealed ulcers, bleeding lesions, tumor, or any other lesion at target magnet deployment site
21. Expected need for MR imaging within the first 2 months after the procedure
22. Any anomaly preventing/contraindicating endoscopic or laparoscopic access and procedures
23. Had surgical or interventional procedure within 30 days prior to procedure
24. Any scheduled surgical or interventional procedure planned within 30 days post- procedure
25. Any stroke/TIA within 6 months prior to consent
26. Requires chronic anticoagulation therapy (except aspirin)
27. Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure
28. Unable to comply with the follow-up schedule and assessments
29. Recent tobacco or nicotine product cessation within < 3 months prior to informed consent
30. Known allergies to the device components or contrast media
31. Limited life expectancy due to terminal disease
32. Currently participating in another clinical research study with an investigational drug or medical device
33. A positive COVID-19 test prior to the study procedure in accordance with local COVID-19 protocol
34. Any condition that, in the investigator's opinion, may preclude completion of follow-up assessments through Day 360 (e.g., a medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, or poor compliance with treatment regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-10-19 (Actual); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Magnet Placement | 1 Day (during study index procedure)
  MagGJ System placement ≥ 90% alignment of magnets
Natural Magnet Passage | Index Procedure through 90 days
  Passage of magnets without surgical re-intervention
Anastomosis Patency | Index Procedure through 90 days
  Confirmed radiologically

CONTACTS AND LOCATIONS:
Locations (1):
- Corporativo Hospital Satelite, Naucalpan, Mexico

IPD SHARING:
Plan to Share IPD: No